CLINICAL TRIAL: NCT05326945
Title: Use of Disposable Sleeve Sheath to Prevent Pathogen Microorganisms Transport From Blood Pressure Cuff
Brief Title: Use of Disposable Cuff Cover to Prevent Carriage of Pathogen Microorganisms Originated by Cuffs
Acronym: DCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aynur KOYUNCU, Principal Investigator, Assist Prof, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HasanKUU
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pathogen Transmission, Vertical; Nosocomial Infection; Cross Infection; Cuff
Keywords: Infection; Nursing; Colonization; Sphygmomanometer Cuff; Pathogen Microorganism
MeSH Terms: conditions — Cross Infection; Infections

STUDY DESIGN:
Intervention Model Description: an experimental clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement without sheath (No Intervention): Sample A: Investigator will take culture from the inside of the BPC, which will contact the patient's right upper arm, wearing sterile gloves, and will remove the gloves.
  B:Investigator will wipe the right upper arm area of the patient with (70% alcohol+2% chlorhexidine) solution in accordance after wearing sterile gloves, wait for 30 seconds and after the alcohol dries investigator will take culture from the patient's right upper arm, wearing a new sterile glove.
  C:investigator will measure ABP on the right upper arm of the patient with the same sterile glove, and after the measurement, the first investigator will take culture from the patient's right upper arm by wearing a new sterile glove, both researchers will remove the gloves.
  D:investigator wore a new sterile glove after ABP measurement and wiped the inside and outside of the BPC with solution, the first investigator would wear a new sterile glove to take culture, both researchers will remove the gloves.
- Sheathed Measurement (Experimental): Sample E: DCC sterile package will be opened the investigator will hold the sphygmomanometer, after investigator wears sterile gloves, DCC will put it cuff of the same cuff. Culture will be taken investigator from the inside of the DCC that will contact the patient's left upper arm, before the ABP measurement, the first investigator will remove the gloves.
  F:Sterile gloves will be worn by the investigator and the left upper arm area of the patient will be wiped with solution before the ABP measurement wait 30 seconds, and after the solution dries, the first investigator will use a new sterile After wearing gloves, he will take a swab culture from the left upper arm region.
  G:The investigator will measure ABP from the patient's left upper arm with the same glove, and after the measurement, the first investigator will take culture from the patient's left upper arm after wearing a new sterile glove.
  Culture results taken from the patients will be compared statistically.
  Interventions: Other: Presence or Absence of a Blood Pressure Cuff Sheath

INTERVENTIONS:
Other: Presence or Absence of a Blood Pressure Cuff Sheath — Monitoring of microorganism transfer from the sphygmomanometer to the patient, from the patient to the sphygmomanometer in case the sheath designed in the research is put on or not before the blood pressure measurement process
  Arms: Sheathed Measurement

SUMMARY:
Introduction: Pathogen Microrganisms (PM) colonized on the Blood Pressure Cuff (BPC) are transported from one patient to another by health professionals, which is leading an increase in Health Care Associated Infections (HCAI). The increase in HCAIs is responsible for the increase in mortality and health expenditures. BPCs cannot be sterilized because they are fixed on blood pressure devices, PMs cannot be completely destroyed by using disinfectant, and disposable BPCs increase health expenditures. A safe and inexpensive method has not yet been found to prevent PMs arising from BPCs that circulate between hospital rooms, moved from patient to patient.

Objective: The aim of this project is to determine the effectiveness of the Disposable Cuff Sleeve (DCS) to be passed over BPCs to prevent the transport of PMs from BPC.

The hypotheses of the study: H1: The use of a DCS is not effective in reducing the transmission of pathogenic microorganisms (number of colonies) originating from the sphygmomanometer cuff to the patient's skin during the arterial blood pressure measurement process.

H2: The use of a disposable cuff cover is effective in reducing the transmission of pathogenic microorganisms (number of colonies) originating from the sphygmomanometer cuff to the patient's skin during the arterial blood pressure measurement process.

Materials and Methods: The study is a clinical study which will be conducted between 28 April- 28 November 2022 in Gaziantep University Hospital. Ethical approval will be obtained before starting the research. The sample of the study will consist of all BPCs (n=100) that are actively used in surgical outpatient clinics, surgical services and surgical intensive care units of Gaziantep Unıversity hospital. Each sphygmomanometer will be used for blood pressure measurement and microorganism determination of a patient. For this purpose, arterial blood pressure (ABP) will be measured from the right and left arm of 116 patients who have been admitted to the outpatient clinics and have accepted to participate in the study. Swabs for a patient's ABP measurement and microorganism determination will take approximately 20-25 minutes. A total of 7 swab cultures will be taken for one sample (one BPC and one patient). Sorting and nomenclature of swab culture will be done as follows:

* Sample A: from the inner part of the BPC in contact with the patient's arm,
* Sample B: upper arm area after wiping with 70% alcohol from upper arm area,
* Sample C: the patient's ABP from the upper arm area after measurement,
* Sample D: After cleaning the inside and outside of BPC with 70% alcohol,
* Sample E: From the inner part of DCS which will contact the patient's arm,
* Sample F: After wiping the upper arm area of the other arm of with 70% alcohol,
* Sample G: will be taken from the upper arm area after the ABP is measured from the other arm.

The swab culture samples taken by the researchers will be delivered to the Microbiology Laboratory of Gaziantep University Hospital within 30 minutes without waiting. The number of PMs and colonies grown in culture samples will be determined according to international standards. The ABP values measured by BPCs (uncoated), DCS' (sheathed) and swab culture results obtained from samples A, B, C, D, E, F, G will be compared statistically. Data analysis will be performed in SPSS 22.0 package program. For statistical significance, p <0.05 will be accepted.

If the H1 hypothesis is confirmed at the end of the study, the use of DSS is proven to be effective in preventing PM transport from BPCs. Prevention of PMs transported from patient to patient with BPCs can lead to a reduction in HCAIs. Reducing HCAIs can reduce mortality and cost increase associated with HCAIs.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old, No fistula, wound or surgical intervention that would prevent blood pressure measurement in both upper arms, Those who have not undergone mastectomy surgery, Not having a diagnosed contagious disease, No tissue ischemia, signs of infection (phlebitis and skin infection), circulation problems, nerve damage, paralysis in the upper arm region, Patients without intravenous or intra-arterial catheters in both arms will be included in the study.

Inclusion Criteria for TAM:

Actively used in surgical outpatient clinics, surgical services, surgical intensive care units for at least one month, Blood pressure devices that measure ABP by wrapping a cuff on the upper arm area, It can be opened completely flat, Sphygmomanometers with the length of the TAM long enough to encircle the upper arm 1.5 times will be included in the research.

Exclusion Criteria:

Patients who want to withdraw from the study at any stage after accepting to participate, TAMs produced for measurement from the lower extremity (leg) or radial artery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-10-28 (Estimated); Study Completion 2022-11-28 (Estimated)

PRIMARY OUTCOMES:
Pathogenic microorganism | Unsheathed blood pressure measurement (without intervention) and sheath blood pressure measurement (with intervention) will be followed up consecutively for each patient. Laboratory results will be sent after 24 hours.
  The number of pathogenic microorganism colonies for each sample

SECONDARY OUTCOMES:
Pathogenic microorganism | Unsheathed blood pressure measurement (without intervention) and sheath blood pressure measurement (with intervention) will be followed up consecutively for each patient. Laboratory results will be sent after 24 hours.
  presence and absence of pathogenic microorganisms

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University Şahinbey Research and Application Hospital, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Clinical Guideline Centre (UK). Infection: Prevention and Control of Healthcare-Associated Infections in Primary and Community Care: Partial Update of NICE Clinical Guideline 2. London: Royal College of Physicians (UK); 2012 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK115271/ PMID 23285500
- [Result] Nguyen LKN, Megiddo I, Howick S. Simulation models for transmission of health care-associated infection: A systematic review. Am J Infect Control. 2020 Jul;48(7):810-821. doi: 10.1016/j.ajic.2019.11.005. Epub 2019 Dec 18. PMID 31862167
- [Result] Suetens C, Latour K, Karki T, Ricchizzi E, Kinross P, Moro ML, Jans B, Hopkins S, Hansen S, Lyytikainen O, Reilly J, Deptula A, Zingg W, Plachouras D, Monnet DL; Healthcare-Associated Infections Prevalence Study Group. Prevalence of healthcare-associated infections, estimated incidence and composite antimicrobial resistance index in acute care hospitals and long-term care facilities: results from two European point prevalence surveys, 2016 to 2017. Euro Surveill. 2018 Nov;23(46):1800516. doi: 10.2807/1560-7917.ES.2018.23.46.1800516. PMID 30458912